CLINICAL TRIAL: NCT06540599
Title: Optimizing Analgesia for Endometrial Biopsy: A Prospective, Randomized Comparative Study
Brief Title: Optimizing Analgesia for Endometrial Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREHes
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2022-03

CONDITIONS: Analgesia
Keywords: endometrial biopsy; intrauterine lidocaine; pain management
MeSH Terms: conditions — Agnosia | interventions — Analgesics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients using intrauterine lidocaine for analgesia (Active Comparator)
  Interventions: Drug: Analgesic
- Patients using oral dexketoprofen for analgesia (Active Comparator)
  Interventions: Drug: Analgesic
- Patients using cervical lidocaine spray for analgesia (Active Comparator)
  Interventions: Drug: Analgesic
- Patients using paracervical block with prilocaine for analgesia (Active Comparator)
  Interventions: Drug: Analgesic

INTERVENTIONS:
Drug: Analgesic — comparing the effectiveness of analgesics in endometrial biopsy

SUMMARY:
Comparison of the effectiveness of intrauterine lidocaine-paracervical block-dexketoprofen tromematol- lidocaine spray in endometrial biopsy analgesia

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-75 needs endometrial biopsy

Exclusion Criteria:

* women with allergies to prilocaine, lidocaine or dexketoprofen trometamol
* women with a history of severe uncontrolled cardiovascular disease, diabetes mellitus, pregnancy, vaginal, cervical, or pelvic infection, cervical cancer, or severe cervical stenosis

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
comparing analgesics in endometrial biopsy using The Visual Analogue Scale (VAS). | 1 hour
  post operative VAS scores will be compared for each drug.The VAS measures pain intensity. The VAS consists of a 10 cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). In this context, higher scores represent worse results.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)